CLINICAL TRIAL: NCT05286411
Title: Evaluation of the Implementation of a Quality Improvement Program Through Morbidity and Mortality Reviews in a Developing Country
Brief Title: Evaluation of the Implementation of a Quality Improvement Program Through Morbidity and Mortality Reviews
Status: Completed | Type: Observational
Sponsor: Moroccan Society of Surgery (Other)
Responsible Party: Principal Investigator, Anass Majbar, Professor MA Majbar, Moroccan Society of Surgery
Other Study IDs: RMM_INO
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Quality Improvement
Keywords: morbidity and mortality reviews; implementation; quality improvement; patient safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Morbidity and mortality reviews represent an opportunity to discuss adverse events and healthcare issues. Aim is to report the first experience of implementing a standardized procedure of morbidity and mortality reviews, and assess its impact on quality improvement.

DETAILED DESCRIPTION:
From July 2019 to December 2019, members of the surgical and intensive care unit departments designed and implemented a regular procedure of morbidity and mortality reviews. Cases of severe postoperative complications after curative resection for digestive cancer were selected to be presented by a surgical resident and discussed in an interdisciplinary conference following a standardized presentation based on an analysis tool adapted from the ALARM framework. Process was assessed by the number of morbidity and mortality reviews held, number and type of recommendations issued and implemented.

Among 13 serious complications during the study period, 10 were discussed. The "Tasks" category was activated in 90% of the cases where lack or misuse of protocols was identified in 90% of the events discussed. Test results availability or accuracy were incarnated in 30% of cases. Poor communication was a contributing factor in 60% of the cases. Written medical records were defective in 40% of the cases. From 16 recommendations for improvement emitted, 87.5% (14/16) were translated into projects and successfully implemented.

Thus, a standardized and regular procedure of morbidity and mortality reviews in a tertiary care facility in a developing country allowed a significant improvement in patient care through quality initiatives implementation. Morbidity and mortality reviews might be a strong tool for the improvement of surgical care particularly for low-mid income countries

ELIGIBILITY:
Inclusion Criteria:

* severe adverse events defined as postoperative morbidity > 3a according to the Clavien Dindo grading system
* within the first 90 postoperative days of surgery
* Cases discussed in a morbidity and mortality review

Exclusion Criteria:

* Cases not discussed in a morbidity mortality review

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent a curative surgical procedure for a digestive cancer in our department during the study period and who presented severe adverse events in 90 post operative day
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Process assessment | one year
  evaluation of the number of MMRs, numbers and categories of identified contributing factors, number and types of recommendations and number and types of implemented recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Oumayma Lahnaoui, MD, Principal Investigator — National Institute of Oncology; Anass Majbar, MD, Study Director — National Institute of Oncology
Locations (1):
- National Institute of Oncology, Rabat, Morocco

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Houssaini K, Lahnaoui O, Souadka A, Majbar MA, Ghanam A, El Ahmadi B, Belkhadir Z, Amrani L, Mohsine R, Benkabbou A. Contributing factors to severe complications after liver resection: an aggregate root cause analysis in 105 consecutive patients. Patient Saf Surg. 2020 Sep 29;14:36. doi: 10.1186/s13037-020-00261-7. eCollection 2020. PMID 33014137
- [Background] Souadka A, Benkabbou A, Al Ahmadi B, Boutayeb S, Majbar MA. Preparing African anticancer centres in the COVID-19 outbreak. Lancet Oncol. 2020 May;21(5):e237. doi: 10.1016/S1470-2045(20)30216-3. Epub 2020 Apr 3. No abstract available. PMID 32251622
- [Background] Souadka A, Majbar MA, Essangri H, Amrani L, Benkabbou A, Mohsine R, Souadka A. Functional outcomes over time following perineal pseudocontinent colostomy reconstruction after abdominoperineal resection for ultralow rectal adenocarcinoma. J Surg Oncol. 2020 Sep;122(4):753-759. doi: 10.1002/jso.26074. Epub 2020 Jun 20. PMID 32563198
- [Background] Majbar MA, Courtot L, Dahbi-Skali L, Rafik A, Jouppe PO, Moussata D, Benkabbou A, Mohsine R, Ouaissi M, Souadka A. Two-step pull-through colo-anal anastomosis aiming to avoid stoma in rectal cancer surgery: A "real life" study in a developing country. J Visc Surg. 2022 Jun;159(3):187-193. doi: 10.1016/j.jviscsurg.2021.04.004. Epub 2021 Jun 4. PMID 34092526